CLINICAL TRIAL: NCT05727514
Title: A Trauma-Informed Music Composition Program Supporting Resilience in Individuals Hospitalized During the COVID-19 Pandemic
Brief Title: Beyond COVID-19: Supporting Resilience With a Trauma-informed Music Composition Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Berklee College of Music (Other)
Responsible Party: Principal Investigator, Nomi Levy-Carrick, MD, MPHIL, Psychiatrist; Vice Chair, Clinical Program, Dept Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021P000904
Record Dates: First submitted 2023-02-08; First posted 2023-02-14 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Problems Related to Life-Management Difficulty

STUDY DESIGN:
Intervention Model Description: case series
Masking Description: participants identity was not disclosed during the program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- enrolled participants (Other): participation in 4-session music composition program with optional viewing of performance at the end
  Interventions: Other: music composition

INTERVENTIONS:
Other: music composition — 4-session music composition program for participants lead by a composer-mentor, includes optional viewing of online string quartet performances of final musical scores

SUMMARY:
This study explores the feasibility and acceptability of a music composition intervention to support resilience in survivors of serious illness hospitalized during the COVID-19 pandemic.

DETAILED DESCRIPTION:
This study explores the feasibility and acceptability of a music composition intervention to support resilience in survivors of serious illness hospitalized during the COVID-19 pandemic. The pandemic introduced widespread trauma for patients facing hospitalization. Therapeutic music interventions have demonstrated positive psychological effects, but none have explored the specific trauma-informed aspects of a composition-mentor program, as well as the specific impact of music composition on resilience-related traits.

Researchers implemented an adapted version of the New York Philharmonic Very Young Composers program (VYC): trained composer-mentors guide participants through four web-based sessions to elicit and develop participants' unique musical ideas into finished compositions. Participants are then invited to view a string quartet performance of their compositions. The Brief Resilience Scale [BRS] and New General Self-Efficacy Scale [NGSE] are administered pre-intervention, post-intervention, and post-performance.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age
* Massachusetts residents
* exhibiting English fluency
* in care with an MGB provider
* admitted as an inpatient for at least 3 days to an MGB hospital between March 15, 2020 and July 21, 2022
* not hospitalized within the month before starting the study.

Exclusion Criteria:

* neuropsychiatric illness impeding participation in the study including suicidality, psychosis, active substance use, and dementia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
New General Self-Efficacy Scale [NGSE] | Data was collected at three time points over 5 months: Pre-Intervention (Baseline: upon enrollment), Post-Intervention (after the final intervention session), and Post-performance (after the final performance).
  The New General Self-Efficacy (NGSE) scale evaluates one's perception of their overall ability to perform successfully in a variety of common scenarios by rating each item from 1-"Strongly Disagree" to 5-"Strongly Agree". Responses were scored by averaging the ratings across items.
  Min possible score: 1 Max possible score: 5
  Min study score: 3.125 Max study score: 5.00
  Higher scores mean a better outcome.
Post-musical composition program questionnaire | Data was collected at one time point, within one week following the final session of the music composition intervention
  Four questions designed for this study elicited open-ended feedback regarding the participant experience of the program: (1) What did you enjoy about this program? (2) What did you find challenging about this program? (3) What did you learn about yourself through this program? (4) Would you recommend this program to other survivors of serious illness?
Post-musical performance program questionnaire | Data was collected at one time point, within two weeks following the end of the music performance
  Four questions designed for this study elicited open-ended feedback regarding the participant experience of listening to their music composition performed by professional musicians: (1) What was it like to hear your composition performed by professional musicians? (2) How did participating in this performance increase the impact of this program overall? (3) Does this program make you feel more confident about being able to be creative in the future? (4) Would you recommend attending the performance as part of this program to other survivors of serious illness?

CONTACTS AND LOCATIONS:
Overall Officials: Nomi Levy-Carrick, MD, MPhil, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No